CLINICAL TRIAL: NCT02681419
Title: Evaluating the Efficacy of Fenestrations in Tube Shunt Implants During the Early Postoperative Period
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Robert Cizik Eye Clinic (Other)
Responsible Party: Principal Investigator, Robert Feldman, Department Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-12-0800
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Needle fenestration (Active Comparator): Needle fenestration
  Interventions: Procedure: Needle fenestration
- Suture wick (Active Comparator): suture wick using 10-0 vicryl
  Interventions: Procedure: Suture wick

INTERVENTIONS:
Procedure: Needle fenestration — This technique creates fenestrations along a nonvalved glaucoma implant (e.g. Baerveldt Glaucoma Implant) anterior to the ligature
  Arms: Needle fenestration
Procedure: Suture wick — This technique places a single 10-vicryl suture wick through the nonvalved glaucoma implant (e.g. Baerveldt Glaucoma Implant) anterior to the ligature
  Arms: Suture wick

SUMMARY:
This study evaluates two different methods of controlling intraocular pressure in nonvalved aqueous tube shunts immediately after implantation; needle fenestrations or a suture wick.

DETAILED DESCRIPTION:
This is a prospective, randomized control study of glaucomatous eye undergoing tube shunt implantation using a nonvalved implant for poorly controlled glaucoma of any type. Eyes scheduled to receive a nonvalved tube shunt implant will be randomized to receive either needle fenestration(s) or a suture wick using a single 10-0 vicryl anterior to the ligature. The operative quadrant will be imaged using anterior-segment optical coherence tomography at pre- and post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Eyes that have poorly controlled glaucoma requiring a tube shunt implantation
* Willingness to participate in the study and sign informed consent

Exclusion Criteria:

* Concurrent surgery except phaco/intraocular lens
* Any abnormality preventing reliable applanation tonometry
* Eyes with exposure limitation (tight lids, deep orbits) that would make performing the anterior segment optical coherence tomography difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with successful control of intraocular pressure | 3 weeks
  Successful control of intraocular pressure is defined as IOP between 5 and 21 mmHg without medications within 3 weeks postop.

SECONDARY OUTCOMES:
Duration of effect on intraocular pressure control | 12 weeks
  The duration of effect is defined as elapsed time from surgery to the time that intraocular pressure (IOP) >5 mmHg or <21 mmHg
Peri-fenestration bleb volume prior to tube opening | 3 weeks
  Bleb volume will be measured by the anterior segment optical coherence tomography (ASOCT)
Peri-fenestration bleb volume after the tube has opened | 12 weeks
  Bleb volume will be measured by the anterior segment optical coherence tomography (ASOCT)
Intraocular pressure after the tube has opened | 12 weeks
  Successful control of intraocular pressure is defined as IOP between 5 and 21 mmHg without medications at 12 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Lauren S. Blieden, MD, Principal Investigator — Robert Cizik Eye Clinic
Locations (1):
- Robert Cizik Eye Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No